CLINICAL TRIAL: NCT01262521
Title: Physiological Effects of Oral Nitrate on Vascular Function
Brief Title: Dietary Nitrate and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Christian Meyer, MD, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Protective dietary nitrate
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: no Medications
Keywords: Dietary nitrate
MeSH Terms: interventions — sodium nitrate; Water

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary nitrate (Experimental): 150 ml tab water with 150 umol/kg sodium-nitrate
  Interventions: Dietary Supplement: Dietary nitrate
- Water (Placebo Comparator): 150 ml Chapelle mineral water
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Dietary nitrate — 150 ml tab water with 150 umol/kg sodium-nitrate
  Other Names: sodium nitrate
  Arms: Dietary nitrate
Dietary Supplement: Water — 150 ml Chapelle mineral water
  Other Names: H2O
  Arms: Water

SUMMARY:
An expanding number of studies suggest a therapeutic role for nitrate and nitrite, most notably in treatment and prevention of cardiovascular disease including ischemia-reperfusion (IR) injury and hypertension. The nutritional aspects of these cardioprotective effects are particularly intriguing since nitrate and nitrite are abundant in our everyday diet.

Whether increasing the circulating pool of nitric oxide and nitrite by dietary nitrate offers a novel mechanistic approach to regulate mobilization of circulating angiogenic cells and thus regenerative processes in cardiovascular medicine is not known. Thus, in the present study, we tested whether oral application of nitrate leads to an enhanced number of circulating angiogenic cells and whether this is associated with an improvement in endothelial function.

DETAILED DESCRIPTION:
Administration of a single dose of nitrate intervention or water alone to healthy volunteers. Before and up to 4 hours (short-term)/6 days (long-term) after ingestion, marker of vascular function are measured in plasma and by using high-resolution ultrasound.

Measurements are taken before and up to 4 h after double blind cross-over per os administration of a single dose of nitrate intervention (150 ml tab water with 150 umol/kg sodium-nitrate) or water control (100 ml Chapelle mineral water) to healthy volunteers. Circulating angiogenic cells are measured as CD34+/KDR+ and CD133+/KDR+ mononuclear cells in blood by flow cytometry and plasma is analyzed for nitrate and nitrite, as well as mobilization markers and cytokines including stromal cell derived factor, vascular endothelial growth factor and stem cell factor. All measurements are performed after >12h overnight fasting.

ELIGIBILITY:
Inclusion Criteria:

* age > 20 years
* refrain from nitrate containing food ingestion during trial

Exclusion Criteria:

* > 36 years
* poor endothelial function
* acute infection
* any chronic heart or pulmonary disease
* arrhythmias
* acute or chronic renal failure
* cardio-vascular risk factors: diabetes mellitus, hypertension, hyperlipidemia
* intake of nutrition supplements (l-arginine, creatinine)

Ages: 21 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Circulating angiogenic cells | 4 hours

SECONDARY OUTCOMES:
Cytokines | 4 hours
Endothelial function | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tienush Rassaf, MD, PhD, Study Chair — University of Duesseldorf; Christian Meyer, MD, Principal Investigator — University of Duesseldorf; Christian Heiss, MD, Principal Investigator — University of Duesseldorf; Malte Kelm, MD, PhD, Study Director — University of Duesseldorf
Locations (1):
- Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Link to the homepage of the Division of Cardiology, Pneumology, and Angiology at the University of Duesseldorf — http://www.uniklinik-duesseldorf.de/kardiologie